CLINICAL TRIAL: NCT03147560
Title: Immunogenicity and Safety Evaluation of Different Sequential Immunization Strategies by Sabin IPV and bOPV in Chinese Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zhejiang Provincial Center for Disease Control and Prevention (Other Government)
Collaborators: China National Biotec Group Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ZJCDC20170508
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Polio
Keywords: Immunogenicity; Safety; Sabin IPV; bOPV
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Experimental): The sequential immunization strategy for group 1 on polio was Sabin IPV+ bOPV + bOPV.
  Interventions: Biological: Sabin IPV+ bOPV+ bOPV
- Group 2 (Experimental): The sequential immunization strategy for group 2 on polio was Sabin IPV + Sabin IPV + bOPV.
  Interventions: Biological: Sabin IPV + Sabin IPV + bOPV
- Group 3 (Experimental): The sequential immunization strategy for group 3 on polio was Sabin IPV + Sabin IPV + Sabin IPV.
  Interventions: Biological: Sabin IPV + Sabin IPV + Sabin IPV

INTERVENTIONS:
Biological: Sabin IPV+ bOPV+ bOPV — Give 3 doses of polio vaccine at 2, 3 and 4 months of age, get 2 blood samples (1.5ml per sample) before the first dose and 28-35 days after the last dose. sIPV was given 0.5ml per dose and bOPV was given 0.1ml per dose.
  Arms: Group 1
Biological: Sabin IPV + Sabin IPV + bOPV — Give 3 doses of polio vaccine at 2, 3 and 4 months of age, get 2 blood samples (1.5ml per sample) before the first dose and 28-35 days after the last dose. sIPV was given 0.5ml per dose and bOPV was given 0.1ml per dose.
  Arms: Group 2
Biological: Sabin IPV + Sabin IPV + Sabin IPV — Give 3 doses of polio vaccine at 2, 3 and 4 months of age, get 2 blood samples (1.5ml per sample) before the first dose and 28-35 days after the last dose. sIPV was given 0.5ml per dose and bOPV was given 0.1ml per dose.
  Arms: Group 3

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of different sequential immunization strategies by Sabin IPV and bOPV in Chinese infants.

ELIGIBILITY:
Inclusion Criteria:

* Parent/legal acceptable representative is willing and able to understand the protocol requirements and provide informed consent.
* Participant is aged ≥ 60 days to ≤ 75 days.
* Participant without preventive inoculation of polio vaccine and previous history of Polio.
* Subject and parent/guardian able to attend all scheduled visits and comply with all trial procedures.
* Body temperature ≤ 37.5℃.

Exclusion Criteria:

* Known allergy to any constituent of the vaccine.
* Known acute illness, severe chronic disease, acute exacerbation of chronic disease and fever.
* Known or suspected impairment of immunologic function, or receipt of immunosuppressive therapy or immunoglobulin since birth.
* Reported the history of allergies, convulsions, epilepsy, mental illness and brain disease and clear serious systemic reaction.
* Known bleeding disorder.
* Receipt of the whole blood, blood plasma or immunoglobulin before the trial vaccination.
* Reported the history of acute illness had need systemic antibiotics or antiviral treatment of infections in the 7 days preceding the trial vaccination.
* An acute illness with or without fever (temperature ≥ 38.0℃) in the 3 days preceding enrollment in the trial.
* Participation in any other intervention clinical trial.
* Any condition which, in the opinion of the investigator, would pose a health risk to the subject or interfere with the vaccine.

Ages: 60 Days to 75 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 528 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
seroconversion rate | seroconversion rate was evaluated 4-5 weeks after the third dose of polio vaccine.
  any positive antibody response in infants who were seronegative prior to their first dose, or at least a fourfold increase in type-specific antibody levels for infants who had pre-existing antibodies.

SECONDARY OUTCOMES:
safety: rate of adverse events | At least 2 active surveillance visits (3 days and 30 days) were required after each vaccination to collect adverse reaction data.
  the rate of adverse events.
neutralizing antibody titer | Blood samples were obtained prior to the first dose and 4-5 weeks after the third dose of polio vaccine.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Chunan Center for Disease Control and Prevention, Hangzhou, Zhejiang
  - Longyou Center for Disease Control and Prevention, Quzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] He H, Wang Y, Deng X, Yue C, Tang X, Li Y, Liu Y, Yin Z, Zhang G, Chen Z, Xie S, Wen N, An Z, Chen Z, Wang H. Immunogenicity of three sequential schedules with Sabin inactivated poliovirus vaccine and bivalent oral poliovirus vaccine in Zhejiang, China: an open-label, randomised, controlled trial. Lancet Infect Dis. 2020 Sep;20(9):1071-1079. doi: 10.1016/S1473-3099(19)30738-8. Epub 2020 May 19. PMID 32442523